CLINICAL TRIAL: NCT01887301
Title: An Open Label, Single-dose, Parallel Group Study to Assess the Pharmacokinetics and Tolerability of a Single Oromucosal Dose of 4 Sprays of Sativex(Containing 10.8 mg Delta-9-tetrahydrocannabinol [THC] and 10 mg Cannabidiol [CBD]) in Patients With Impaired Hepatic Function and Healthy Subjects With Normal Hepatic Function.
Brief Title: Assessment of the Single Dose Pharmacokinetics and Tolerability of Sativex in Patients With Impaired Hepatic Function and Healthy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWCP10114
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: mild hepatic impairment (Active Comparator): Mild hepatic impairment: eight patients of Child-Pugh Grade A (Score 5-6). All patients received Sativex treatment.
  Interventions: Drug: Sativex
- Group 2: Moderate hepatic impairment (Active Comparator): Moderate hepatic impairment: eight patients of Child-Pugh Grade B (Score 7-9). All patients received Sativex treatment.
  Interventions: Drug: Sativex
- Group 3: Pugh Grade B (Score 7-9). (Experimental): Severe hepatic impairment: eight patients of Child-Pugh Grade C (Score 10-15). All patients received Sativex treatment.
  Interventions: Drug: Sativex
- Group 4: Control group (Active Comparator): Control Group: eight healthy subjects matched with respect to age (±10 years), weight (±10% body mass index [BMI]) and sex to the severe or most severe evaluable patients. All patients received Sativex treatment.
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Patients receive four sprays (each 100 uL) of Sativex to the oral mucosa, which contain 10.8 mg THC and 10 mg CBD in total.
  Other Names: Nabiximols; GW1000-02; THC/CBD spray

SUMMARY:
A Phase I open-label study to evaluate the pharmacokinetics (what the body does to a drug), safety and tolerability of a single dose of Sativex (containing 10.8 mg tetrahydrocannabinol [THC] and 10 mg cannabidiol [CBD]) in healthy patients and those with hepatic (liver) function impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 18 years or above.
* Subject is willing and able to give informed consent for participation in the study (see Section 14.2).
* Male or female subjects.
* All females must have negative pregnancy test results at screening and baseline.
* Vital signs (after five minutes resting measured in the supine position) must be within the following ranges:
* Body temperature between 35.0-37.5 °C
* Systolic blood pressure, 90-150 mmHg
* Diastolic blood pressure, 60-90 mmHg
* Pulse rate, 40-99 beats per minute (bpm) Blood pressure and pulse will be taken again in a standing position. After two minutes standing, there shall be no more than a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure, associated with clinical manifestation of postural hypotension.
* Subjects must weigh at least 50 kg and have a BMI between 19 and 42 kg/m2 to participate in this study.
* Patients with impaired hepatic function must be compliantly on a stable dose of medication and/or treatment regimen (in the opinion of the investigator) for at least 4 weeks prior to the dosing day with no foreseeable plans for change.
* Subject is able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing and able to communicate well with the Investigator.
* Subject is willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
* Subject is willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Groups 1 and 2 (mild and moderate hepatic impairment)

* Clinical features consistent with a confirmed clinical diagnosis of mild and moderate liver impairment.
* Child-Pugh clinical assessment score consistent with degree of hepatic impairment.
* Clinical evidence of stable hepatic impairment, defined as no clinically significant change in disease status within the last 30 days, as documented by the patients' recent medical history.
* Otherwise considered healthy in general as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at screening.
* Platelet count > 50,000 X 109/L at screening and baseline.
* Willing to maintain a stable dose of any, not prohibited, medication throughout the study.

Group 3 (severe hepatic impairment)

* Patients presenting at least one clinical sign consistent with a clinical diagnosis of severe liver impairment.
* Child-Pugh clinical assessment score consistent with degree of hepatic impairment.
* Platelet count > 30,000 X 109/L at screening and baseline.
* Willing to maintain a stable dose of any, not prohibited, medication throughout the study.

Group 4 (healthy controls)

* In good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at screening.
* Healthy male or female subjects, matched with respect to age (±10 years), weight (±10% BMI) and sex to the severe or most severe evaluable patients.
* No clinical evidence of liver disease or liver injury as indicated by clinically significant abnormal liver function tests such as aspartate aminotransferase, alanine aminotransferase, γ-glutamyl-transpeptidase, alkaline phosphatase, or serum bilirubin two times above the upper limit of the normal range.

Exclusion Criteria:

* Donation or loss of 400 mL or more of blood within eight weeks prior to dosing.
* Significant concomitant illness within the two weeks prior to dosing.
* Resting heart rate <40 bpm.
* History of autonomic dysfunction.
* History of clinically significant drug allergy; a known hypersensitivity to the study drug or drugs similar to the study drug.
* Any surgical or medical condition (other than hepatic impairment) which might significantly alter the absorption, distribution, metabolism or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
* Any history of significant bleeding and haemorrhagic tendencies. However, subjects with a history of bleeding tendencies secondary to hepatic impairment will be excluded based on Principal Investigators' discretion.
* History of immunocompromisation, including known history of human immunodeficiency virus seropositivity.
* History of drug abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Unwilling to abstain from alcohol during this study.
* Currently receiving a prohibited or restricted medication and unwilling to stop or comply with restriction for 14 days prior to the screening visit and for the duration of the study.
* Currently using or has used cannabis, cannabinoid-based medications (e.g. Marinol, Nabilone, Cannador), or Acomplia (rimonabant) or taranabant within 30 days of study entry and unwilling to abstain for the duration of the study.
* A known or suspected history or family history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with underlying condition.
* A history of uncontrolled epilepsy as evidenced by one or more seizures in the last 12 months.
* Significant cardiac disease, e.g. has experienced myocardial infarction (MI) (if the screening ECG reveals patterns consistent with a MI and the date of the event cannot be determined, then the subject can enter the study at the discretion of the Investigator and/or local medical monitor) or clinically relevant cardiac dysfunction within the last six months, or any of the following within the last six months:
* had a coronary artery bypass surgery or percutaneous coronary intervention,
* has unstable angina or has had stroke,
* unstable heart insufficiency (New York Heart Association grade III-IV),
* has a cardiac disorder that, in the opinion of the Investigator, would put the subject at risk of a clinically relevant arrhythmia or MI, or has a secondary or tertiary atrioventricular block.
* Had liver surgery (including transplantation) within the last six months.
* Has significant renal disease or significantly impaired renal function with a creatinine clearance below 50 mL/min for Group 1 and 2, or below 40 mL/min for Group 3.
* Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception, for example, oral contraception, double barrier or intra-uterine device, during the study and for three months thereafter (however, a male condom should not be used in conjunction with a female condom as this may not prove effective).
* Female subject who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Any clinically significant abnormal findings in physical or oral examination, ECG or laboratory evaluations (not consistent with known clinical disease) which, in the opinion of the Investigator, may put the subject at risk, influence the result of the study, or the subjects' ability to participate in the study.
* Subjects who are unwilling to abstain from smoking from midnight on Day -1 to four hours post dose Day 1.
* Subjects who consume more than five caffeinated beverages per day (e.g. five cups of tea or coffee or cans of cola) or who are unwilling to abstain from consumption of caffeine-containing food and beverages throughout the period of in-patient confinement.
* Unwilling to abstain from donation of blood during the study.
* Travel outside the country of residence planned during the study.
* Subjects previously enrolled into this study.
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal product (IMP).
* Subjects who have received an IMP within 30 days or five times the half-life of the IMP (whichever is greater) prior to the screening visit.

Groups 1, 2, and 3 (hepatic impairment)

* Symptoms or history of Stage III or worse degree of encephalopathy.
* Clinical evidence of severe ascites.
* Any evidence of acute progressive liver disease.
* Patients with clinically abnormal prothrombin time will be excluded based on the Principal Investigators' discretion.

Group 4 (healthy controls)

* A positive Hepatitis B surface antigen or Hepatitis C test result.
* History of alcohol abuse within the 12 months prior to dosing or evidence of such abuse, as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Use of any prescription medication within 14 days prior to dosing except for hormonal contraceptives.
* Use of over-the-counter medications or vitamins within 14 days prior to dosing (except for the occasional use of paracetamol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic analysis - Unbound maximum plasma concentration (Cmax(u)) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of unbound THC, CBD, 11-hydroxy-THC (11-OH-THC), 6-hydroxy-CBD (6-OH-CBD) and 7-hydroxy-CBD (7-OH-CBD).
Pharmacokinetic analysis - Unbound area under the concentration-time curve calculated to the last observable concentration at time t (AUC0-t(u)) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of unbound THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.
Pharmacokinetic analysis - Unbound Area under the concentration-time curve from time zero to infinity (AUC0-inf(u)) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of unbound THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.

SECONDARY OUTCOMES:
Pharmacokinetic analysis - Maximum (peak) plasma concentration (Cmax) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.
Pharmacokinetic analysis - Area under the concentration-time curve calculated to the last observable concentration at time t (AUC0-t) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.
Pharmacokinetic analysis - Area under the concentration-time curve from time zero to infinity (AUC0-inf) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.
Pharmacokinetic analysis - Half-Life (t1/2) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.
Pharmacokinetic analysis - time to peak concentration (Tmax) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of THC, CBD, 11-OH-THC, 6-OH-CBD and 7-OH-CBD.
Pharmacokinetic analysis - Apparent unbound clearance of drug from plasma (CL(u)/F) of Sativex® in healthy patients and in patients with hepatic impairment | Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose.
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For pharmacokinetic (PK) assessments, blood will be drawn from each patient into a five mL lithium-heparinised tube at the following intervals (±five min): Pre-dose (0),0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 11, 24, 36 and 48 hours post dose. Collected blood samples will be used to confirm correct dosing, and to provide information about the plasma concentrations of THC, CBD.
Incidence of adverse events during the study | Days 1-7
  Any adverse changes in the patients' medical condition following completion of the consent form were recorded on the case report forma as adverse events. The number of patients who experienced an adverse event is presented.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Clinical Pharmacology of Miami, Inc., Miami, Florida